CLINICAL TRIAL: NCT06764147
Title: Phase 1 Pharmacokinetic Study of Methoxyethyl Etomidate Hydrochloride for Injection With a Single Dose in Elderly Subjects
Brief Title: Safety and Pharmacokinetics/ Pharmacodynamics of Methoxyethyl Etomidate Hydrochloride in Healthy Elderly Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ahon Pharmaceutical Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ET-26-HCL-CP-005
Record Dates: First submitted 2024-12-19; First posted 2025-01-08 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Healthy Elderly Subjects
MeSH Terms: interventions — ET-26 compound

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non-elderly group (Experimental): aged 18-64 years (including boundary value)
  Interventions: Drug: ET-26HCl
- Elderly group (Experimental): aged ≥65 years old, of which no less than 3 cases were ≥75 years old
  Interventions: Drug: ET-26HCl

INTERVENTIONS:
Drug: ET-26HCl — The dose is 0.8 mg/kg, single dose, Infusion time was 60s ± 5s.

SUMMARY:
16 subjects were divided into two groups: One group consisted of healthy non-elderly subjects aged 18-64 years (including boundary value). The other group was healthy elderly subjects, aged ≥65 years old, of which no less than 3 cases were ≥75 years old, with 8 subjects in each group.Healthy non-elderly subjects will be included as matched control subjects. The gender of healthy non-elderly subjects was consistent with that of healthy elderly subjects. The mean body weight of the healthy non-elderly subjects was within the range of the mean body weight of the healthy elderly subjects ±10 kg.

All patients received a single intravenous injection of 0.8mg/kg ET-26. To evaluate the pharmacokinetic characteristics of ET-26 and provide guidance for the clinical application of ET-26-hcl.

ELIGIBILITY:
Inclusion Criteria:

1. healthy adult male and female subjects aged ≥18 years;
2. Body weight: body mass index (BMI) between 19.0 and 28.0 kg/m2 (including the cut-off value), with a body weight of at least 50 kg for male subjects and 45 kg for female subjects;
3. Blood pressure of healthy subjects should be between 90-139/60-89 mmHg, heart rate and pulse should be between 55-100 beats/min
4. The subjects had good communication with the investigators, signed the informed consent form voluntarily, and were able to complete the trial according to the protocol.

Exclusion Criteria:

-

Auxiliary examination:

1. If the results of physical examination, vital signs, color Doppler echocardiography (only for healthy elderly subjects), cortisol test, laboratory tests (blood routine, blood biochemistry, coagulation function, urine routine) and 12-lead electrocardiogram were abnormal and clinically significant by investigator evaluation;
2. potentially difficult airway (modified Mallampati score III-IV);
3. hepatitis B surface antigen, hepatitis C antibody, HIV antibody or syphilis antibody positive;

   Medication history:
4. use of any drugs that inhibit or induce hepatic drug-metabolizing enzymes within 30 days before screening;
5. use of any prescribed medication within 14 days before dosing;
6. use of over-the-counter drugs, Chinese herbal medicines or food supplements such as vitamins and calcium supplements within 7 days before administration;

   History of disease and surgery:
7. have a history of any clinically serious diseases or diseases or conditions considered by the investigators to be likely to affect the results of the trial, including but not limited to a history of circulatory, respiratory, endocrine, nervous, digestive, urinary, or hematologic, immune, psychiatric, or metabolic diseases;
8. patients with a history of adrenal insufficiency, adrenal tumors, or hereditary heme biosynthesis disorders;
9. patients who underwent any surgery within 6 months before screening;
10. Allergic constitution, such as known allergic history to two or more substances; Or who, as judged by the investigator, may be allergic to the trial drug or its excipients;

    Living habits:
11. binge drinking or regular drinking in the 6 months before screening, i.e. more than 14 units of alcohol per week (1 unit =360 mL of beer or 45 mL of 40% spirits or 150 mL of wine); Or with a positive alcohol breath test at baseline;
12. if they smoked more than 5 cigarettes per day in the 3 months before screening or could not quit smoking during the study;
13. with drug abuse or drug abuse history in the past three months; Or the baseline urine drug test was positive;
14. habitual consumption of grapefruit juice or excessive tea, coffee and/or caffeinated beverages and inability to quit during the trial;

    Others:
15. those who have difficulty in blood collection, can not tolerate venipuncture, and can not tolerate arterial blood collection (e.g. Allen's test positive);
16. participated in any other clinical trial (including drug and device clinical trial) within 3 months before screening;
17. vaccinated within 1 month before screening or planned to be vaccinated during the trial period;
18. pregnant or lactating women;
19. those who planned to give birth or donate sperm during the trial and half a year after the completion of the trial, or those who did not agree that the subjects and their spouses should take strict contraceptive measures during the trial and half a year after the completion of the trial;
20. had blood loss or donation >400 mL within 3 months before screening, or received blood transfusion within 1 month;
21. subjects with any factors considered by the investigator to be ineligible for the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2023-12-25 (Actual); Primary Completion 2024-02-02 (Actual); Study Completion 2024-02-02 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameters | up to 24 hours after infusion
  Cmax
Pharmacokinetic parameters | up to 6 hours after infusion
  Tmax
Pharmacokinetic parameters | up to 12 hours after infusion
  T1/2
Pharmacokinetic parameters | immediately after infusion to 24 hours after infusion
  AUC0-t

SECONDARY OUTCOMES:
Pharmacodynamic indicators | MOAA/S score was measured within 60 minutes before administration, was performed every 1 minute±5second within 5minutes of administration and every 2minutes ±30seconds after 5minutes of administration
  modified observer's assessment of alert（MOAA/S） score: The lowest score was 0, indicating full anesthetic sedation, and the highest score was 5, indicating full consciousness
Pharmacodynamic indicators | BIS score was measured within 60 minutes before administration as baseline value,was performed every 1 minute±5second within 5minutes of administration and every 2minutes±30seconds after 5minutes of administration
  bispectral index: BIS values range from 0 to 100, with higher values indicating more wakefulness and lower values indicating more severe cortical inhibition.
Pharmacodynamic indicators：Eyelash reflex | every 1 minute± 5seconds during the first 5minutes of administration and every 2minutes ±30seconds after 5minutes of administration
  When the anesthesiologist touches the eyelashes with the anterior fibers of the cotton swab, it can cause the blink of the examined person, that is, there is an eyelash reflex. If the reaction disappears, the depth of anesthesia is judged to reach the degree of loss of consciousness

CONTACTS AND LOCATIONS:
Overall Officials: Wei Zhao, Pharmaciae Doctor, Principal Investigator — The First Affiliated Hospital of Shandong First Medical University (Qianfoshan Hospital of Shandong Province)
Locations (1):
- The First Affiliated Hospital of Shandong First Medical University (Qianfoshan Hospital of Shandong Province), Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: Undecided